CLINICAL TRIAL: NCT01341639
Title: A Phase III Randomized, Double-Blind, Active-Comparator Controlled Clinical Trial to Study the Safety, Tolerability, and Immunogenicity of V419 in Healthy Infants When Given at 2, 3, 4, and 12 Months (V419-007-03)
Brief Title: Safety, Tolerability, and Immunogenicity of V419 in Healthy Infants When Given at 2, 3, 4 and 12 Months (V419-007)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MCM Vaccines B.V. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V419-007; 2010-021490-37 (EudraCT Number)
Record Dates: First submitted 2011-04-22; First posted 2011-04-26 (Estimated); Results first posted 2019-04-10 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Bacterial Infections; Virus Diseases
Keywords: combination vaccine; diphtheria; pertussis; tetanus; hepatitis B; Hep B; Haemophilus influenzae b; Hib; polio; poliovirus
MeSH Terms: conditions — Bacterial Infections; Virus Diseases; Diphtheria; Whooping Cough; Tetanus; Hepatitis B; Haemophilus Infections; Poliomyelitis | interventions — RotaTeq; 13-valent pneumococcal vaccine; measles, mumps, rubella, varicella vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PR5I (Experimental): V419 + RotaTeq + Prevenar 13 + ProQuad
  Interventions: Biological: V419; Biological: RotaTeq; Biological: Prevenar 13; Biological: ProQuad™
- INFANRIX™ hexa (Active Comparator): INFANRIX™ hexa + RotaTeq + Prevenar 13 + ProQuad
  Interventions: Biological: INFANRIX™ hexa; Biological: RotaTeq; Biological: Prevenar 13; Biological: ProQuad™

INTERVENTIONS:
Biological: V419 — V419 (Diphtheria and Tetanus Toxoids and Acellular Pertussis Adsorbed, Inactivated Poliovirus, Haemophilus b Conjugate [Meningococcal Outer Membrane Protein Complex], and Hepatitis B [Recombinant] Vaccine) 0.5 mL intramuscular injection at 2, 3, 4, and 12 months of age.
  Arms: PR5I
Biological: INFANRIX™ hexa — INFANRIX™ hexa 0.5 mL intramuscular injection at 2, 3, 4, and 12 months of age.
  Arms: INFANRIX™ hexa
Biological: RotaTeq — RotaTeq (pentavalent combination live vaccine of 5 human-bovine reassortant rotavirus strains) 2 mL oral dose at 2, 3, and 4 months of age
Biological: Prevenar 13 — Prevenar 13 0.5 mL intramuscular injection at 2, 3, 4,and 13 months of age
Biological: ProQuad™ — ProQuad™ 0.5 mL subcutaneous injection at 12 and 13 months of age

SUMMARY:
This study will determine whether participants who receive the vaccine V419 at 2, 3, 4, and 12 months of age have an acceptable immune response to the vaccine. The study will also determine whether the immune response to V419 is similar to that of participants who receive a licensed vaccine control.

ELIGIBILITY:
Inclusion Criteria

* Healthy infants able to attend all study visits
* Parent(s)/legal representative able to read, understand, and complete study questionnaires

Exclusion Criteria

* History of congenital or acquired immunodeficiency
* Received or is expected to receive immunosuppressive agents or systemic immunomodulatory steroids
* History of leukemia, lymphoma, malignant melanoma, or myeloproliferative disorder
* Hypersensitivity to any of the vaccine components or history of a life-threatening reaction to a vaccine containing the same substances as the study vaccines or concomitant study vaccines
* Has any chronic illness that could interfere with study conduct or completion
* Received any immune globulin, blood, or blood-derived products since birth
* Received a dose of hepatitis B vaccine prior to the study
* Vaccinated with any acellular pertussis or whole cell pertussis based combination vaccines, Haemophilus influenzae type b conjugate, poliovirus, pneumococcal conjugate or pneumococcal polysaccharide, rotavirus, measles, mumps, rubella, or varicella vaccines, or any combination thereof
* Fever within 24 hours prior to enrollment
* Received any non-study vaccine within 30 days prior to enrollment, except for inactivated influenza vaccine, which is permitted 14 days or more prior to enrollment
* Has a coagulation disorder
* Has developmental delay or neurological disorder
* Participant or his/her mother has a medical history of hepatitis B surface antigen (HBsAg) seropositivity
* History of measles, mumps, rubella, varicella, Haemophilus influenzae type B, hepatitis B, diphtheria, tetanus, pertussis, rotavirus, invasive pneumococcal, or poliomyelitis infection

Ages: 46 Days to 74 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1250 (Actual)
Dates: Start 2011-05-26 (Actual); Primary Completion 2013-03-13 (Actual); Study Completion 2013-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Vesikari T, Becker T, Vertruyen AF, Poschet K, Flores SA, Pagnoni MF, Xu J, Liu GF, Stek JE, Boisnard F, Thomas S, Ziani E, Lee AW. A Phase III Randomized, Double-blind, Clinical Trial of an Investigational Hexavalent Vaccine Given at Two, Three, Four and Twelve Months. Pediatr Infect Dis J. 2017 Feb;36(2):209-215. doi: 10.1097/INF.0000000000001406. PMID 27846055

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy infants 46 to 74 days old were enrolled in this study.
Groups:
- PR5I: The PR5I group received V419, Prevenar 13™, and RotaTeq™ at 2, 3, and 4 months; followed by V419 and ProQuad™ at 12 months, and Prevenar 13™ and ProQuad™ at 13 months.
- INFANRIX™ Hexa: The INFANRIX™ hexa group received INFANRIX™ hexa, Prevenar 13™, and RotaTeq™ at 2, 3, and 4 months; followed by INFANRIX™ hexa and ProQuad™ at 12 months; and Prevenar 13™ and ProQuad™ at 13 months.
Period: Infant Series
Arm/Group | PR5I | INFANRIX™ Hexa
Started (All Randomized Participants) | 628 | 622
Site 0048 Excluded (Participants from Site 0048 were excluded from all analyses due to major findings in study conduct.) | 611 | 606
Treated | 610 | 605
Completed | 599 | 590
Not Completed | 29 | 32
Not completed — Protocol Violation | 1 | 0
Not completed — Not Vaccinated | 0 | 1
Not completed — Adverse Event | 0 | 5
Not completed — Withdrawal by Subject | 11 | 8
Not completed — Lost to Follow-up | 0 | 2
Not completed — Site 0048 Participants | 17 | 16
Period: Interim Period
Arm/Group | PR5I | INFANRIX™ Hexa
Started | 599 | 590
Completed | 591 | 581
Not Completed | 8 | 9
Not completed — Withdrawal by Subject | 6 | 7
Not completed — Lost to Follow-up | 2 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 0 | 1
Period: Toddler Dose
Arm/Group | PR5I | INFANRIX™ Hexa
Started | 590 (One participant randomized to the PR5I group mistakenly received INFANRIX™ hexa instead) | 582 (One participant randomized to the PR5I group mistakenly received INFANRIX™ hexa instead)
Completed | 539 | 548
Not Completed | 51 | 34
Period: Post-Treatment
Arm/Group | PR5I | INFANRIX™ Hexa
Started | 539 | 548
Completed | 539 | 545
Not Completed | 0 | 3
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants excluding participants from site 0048.
Groups:
- Total: Total of all reporting groups
Arm/Group | PR5I | INFANRIX™ Hexa | Total
Number analyzed (Participants) | 611 | 606 | 1217
Age, Continuous [Mean (Standard Deviation); unit: Days] | 61.4 (6.9) | 61.5 (6.9) | 61.5 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 291 | 290 | 581
  Male | 320 | 316 | 636

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Vaccinated With PR5I With Acceptable Antibody (Ab) Response to Haemophilus Influenzae Type b, Diphtheria, Tetanus, and Poliovirus Types 1, 2 & 3, at 5 Months
Description: Antibody titres in the PR5I group were measured by Radioimmunoassay (RIA) for Haemophilus influenzae type b (PRP), Micrometabolic inhibition test (MIT) for diphtheria & poliovirus, and Enzyme-Linked Immunosorbent Assay (ELISA) for tetanus. Percentage of participants with an Ab titre ≥0.15 μg/mL for Haemophilus influenzae type b (Hib) (polyribosylribitol phosphate, PRP); ≥0.01 IU/mL; for diphtheria & tetanus; ≥8 (1/dil) for inactivated poliovirus types 1, 2 & 3 (IPV1, 2 & 3) are reported. 95% confidence interval (CI) were calculated based on the exact binomial method by Clopper and Pearson. The immune response to PR5I vaccine was considered as acceptable if the lower bounds of the 2-sided 95% CI for the response rates were greater than the predetermined lower CI limits for PRP, diphtheria (80%), tetanus (90%), and IPV1, 2 & 3 (90%).
Time Frame: One month after post-dose 3 of PRI5 (5 months old)
Population: All participants in the PR5I group who met inclusion criteria, were not protocol violators, received vaccinations within acceptable day ranges, and who had serology results within revised windows (RW) of Days 28 to 51 Post-Dose 3. Participants from site 0048 were excluded. Participants in the INFANRIX™ hexa group were not analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PR5I
Number analyzed (Participants) | 550
Percentage of participants
  Anti-PRP ≥0.15 μg/mL | 98.36 [96.92 to 99.25]
  Anti-Diphtheria ≥0.01 IU/mL: number analyzed (Participants) | 542
  Anti-Diphtheria ≥0.01 IU/mL | 99.82 [98.98 to 100]
  Anti-Tetanus ≥0.01 IU/mL: number analyzed (Participants) | 538
  Anti-Tetanus ≥0.01 IU/mL | 100 [99.32 to 100]
  Anti-IPV1 ≥8 (1/dil): number analyzed (Participants) | 547
  Anti-IPV1 ≥8 (1/dil) | 100 [99.33 to 100]
  Anti-IPV2 ≥8 (1/dil): number analyzed (Participants) | 547
  Anti-IPV2 ≥8 (1/dil) | 99.82 [98.99 to 100]
  Anti-IPV3 ≥8 (1/dil): number analyzed (Participants) | 545
  Anti-IPV3 ≥8 (1/dil) | 100 [99.33 to 100]

2. Primary Outcome: Percentage of Participants Vaccinated With PR5I With Acceptable Ab Response or Seroresponse Rates to All Antigens Contained in the PR5I Vaccine One Month After the Toddler Dose at 13 Months
Description: Antibody titres in the PR5I group were measured by RIA for PRP, MIT for diphtheria & poliovirus, enhanced Chemiluminescence assay (ECi)) for Hepatitis B surface antigen (HBsAg) and ELISA for tetanus, Pertussis toxoid (PT), Filamentous haemagglutinin (FHA), Fimbriae types 2 & 3 (FIM) & Pertactin (PRN). Percentage of participants with an Ab titre ≥1.0 μg/mL for Hib (PRP); ≥0.1 IU/mL; for diphtheria & tetanus; ≥10 mIU/mL HBsAg; ≥8 (1/dil) for IPV1, 2 & 3, and seroresponse to PT, FHA, FIM and PRN are reported. 95% confidence interval (CI) were calculated based on the exact binomial method by Clopper and Pearson. The immune response to PR5I vaccine was considered as acceptable if the lower bounds of the 2-sided 95% CI for the response rates were greater than the lower CI limits for PRP, PT, FHA, FIM, and PRN (75%); Diphtheria (80%); HBsAG, IPV 1, 2, 3 (90%).
Time Frame: One month after Toddler dose of PRI5 (13 months old)
Population: All participants in the PR5I group who met inclusion criteria, were not protocol violators, received vaccinations within acceptable day ranges, and who had serology results within RW of Days 28 to 51 Post-Toddler dose. Participants from site 0048 were excluded. Participants in the INFANRIX™ hexa group were not analyzed for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PR5I
Number analyzed (Participants) | 551
Percentage of participants
  Anti-PRP ≥1.0 μg/mL: number analyzed (Participants) | 439
  Anti-PRP ≥1.0 μg/mL | 94.99 [92.51 to 96.83]
  Anti-Diphtheria ≥0.1 IU/mL: number analyzed (Participants) | 531
  Anti-Diphtheria ≥0.1 IU/mL | 99.81 [98.96 to 100]
  Anti-Tetanus ≥0.1 IU/mL: number analyzed (Participants) | 538
  Anti-Tetanus ≥0.1 IU/mL | 100 [99.3 to 100]
  Anti-IPV1 ≥8 (1/dil): number analyzed (Participants) | 538
  Anti-IPV1 ≥8 (1/dil) | 99.81 [98.97 to 100]
  Anti-IPV2 ≥8 (1/dil): number analyzed (Participants) | 538
  Anti-IPV2 ≥8 (1/dil) | 100 [99.32 to 100]
  Anti-IPV3 ≥8 (1/dil): number analyzed (Participants) | 541
  Anti-IPV3 ≥8 (1/dil) | 100 [99.32 to 100]
  Anti-HBsAg ≥10 mIU/mL | 99.64 [98.7 to 99.96]
  Anti-PT seroresponse: number analyzed (Participants) | 543
  Anti-PT seroresponse | 99.82 [98.98 to 100]
  Anti-FHA seroresponse: number analyzed (Participants) | 542
  Anti-FHA seroresponse | 97.23 [95.48 to 98.44]
  Anti-FIM seroresponse: number analyzed (Participants) | 508
  Anti-FIM seroresponse | 99.61 [98.59 to 99.95]
  Anti-PRN seroresponse: number analyzed (Participants) | 543
  Anti-PRN seroresponse | 98.9 [97.61 to 99.59]

3. Primary Outcome: Percentage of Participants Vaccinated With PR5I Compared With INFANRIX™ Hexa With Acceptable Ab Response to Haemophilus Influenzae Type b, Diphtheria, Tetanus, and Poliovirus Types 1, 2 & 3, at 5 Months
Description: Antibody titres were measured by RIA for PRP, MIT for diphtheria & poliovirus, and ELISA for tetanus. Percentage of participants with an Ab titre ≥0.15 μg/mL for Hib) (PRP); ≥0.01 IU/mL; for diphtheria & tetanus; ≥8 (1/dil) for inactivated poliovirus types 1, 2 & 3 (IPV1, 2 & 3) are reported. The estimated response rates are based on the method by Miettinen and Nurminen stratified by country.
Time Frame: One month after post-dose 3 of PRI5 (5 months old)
Population: All participants who met inclusion criteria, were not protocol violators, received vaccinations within acceptable day ranges, and who had serology results within RW of Days 28 to 51 Post-Dose 3. Participants from site 0048 were excluded.
Measure: Number; unit: Percentage of participants
Arm/Group | PR5I | INFANRIX™ Hexa
Number analyzed (Participants) | 550 | 530
Percentage of participants
  Anti-PRP ≥0.15 μg/mL: number analyzed (Participants) | 550 | 521
  Anti-PRP ≥0.15 μg/mL | 98.36 | 86.99
  Anti-Diphtheria ≥0.01 IU/mL: number analyzed (Participants) | 542 | 517
  Anti-Diphtheria ≥0.01 IU/mL | 99.81 | 99.81
  Anti-Tetanus ≥0.01 IU/mL: number analyzed (Participants) | 538 | 519
  Anti-Tetanus ≥0.01 IU/mL | 100 | 100
  Anti-IPV1 ≥8 (1/dil): number analyzed (Participants) | 547 | 528
  Anti-IPV1 ≥8 (1/dil) | 100 | 99.81
  Anti-IPV2 ≥8 (1/dil): number analyzed (Participants) | 547 | 530
  Anti-IPV2 ≥8 (1/dil) | 99.82 | 99.62
  Anti-IPV3 ≥8 (1/dil): number analyzed (Participants) | 545 | 525
  Anti-IPV3 ≥8 (1/dil) | 100 | 100
Statistical Analysis 1: Comparison: PR5I vs INFANRIX™ Hexa; Difference in percentages: Non-inferiority for PRP; Test type: Non-Inferiority — If the lower bound of the 95% CI was greater than -10% (non-inferiority margin), it was concluded that PR5I group response rate was non-inferior to INFANRIX hexa group response rate; p < 0.001, Miettinen & Nurminen — 1-sided; Difference in percentages = 11.37, 95% CI 2-sided [8.44 to 14.68] — If the lower bound of the 95% CI was greater than -10% (non-inferiority margin), it was concluded that PR5I group response rate was non-inferior to INFANRIX hexa group response rate; PR5I minus INFANRIX™ hexa
Statistical Analysis 2: Comparison: PR5I vs INFANRIX™ Hexa; Difference in percentages: Non-inferiority for Diphtheria; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; p < 0.001, Miettinen & Nurminen — 1-sided; Difference in percentages = 0, 95% CI 2-sided [-0.95 to 0.96] — [estimate comment as in outcome 3, analysis 1]; PR5I minus INFANRIX™ hexa
Statistical Analysis 3: Comparison: PR5I vs INFANRIX™ Hexa; Difference in percentages: Non-inferiority for Tetanus; Test type: Non-Inferiority — If the lower bound of the 95% CI was greater than -5% (non-inferiority margin), it was concluded that PR5I group response rate was non-inferior to INFANRIX hexa group response rate; p < 0.001, Miettinen & Nurminen; Difference in percentages = 0, 95% CI 2-sided [-0.71 to 0.74] — If the lower bound of the 95% CI was greater than -5% (non-inferiority margin), it was concluded that PR5I group response rate was non-inferior to INFANRIX hexa group response rate; PR5I minus INFANRIX™ hexa
Statistical Analysis 4: Comparison: PR5I vs INFANRIX™ Hexa; Difference in percentages: Non-inferiority for IPV1; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 3]; p < 0.001, Miettinen & Nurminen — 1-sided; Difference in percentages = 0.19, 95% CI 2-sided [-0.51 to 1.07] — [estimate comment as in outcome 3, analysis 3]; PR5I minus INFANRIX™ hexa
Statistical Analysis 5: Comparison: PR5I vs INFANRIX™ Hexa; Difference in percentages: Non-inferiority for IPV2; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 3]; p < 0.001, Miettinen & Nurminen — 1-sided; Difference in percentages = 0.19, 95% CI 2-sided [-0.69 to 1.21] — [estimate comment as in outcome 3, analysis 3]; PR5I minus INFANRIX™ hexa
Statistical Analysis 6: Comparison: PR5I vs INFANRIX™ Hexa; Difference in percentages: Non-inferiority for IPV3; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 3]; p < 0.001, Miettinen & Nurminen — 1-sided; Difference in percentages = 0, 95% CI 2-sided [-0.7 to 0.73] — [estimate comment as in outcome 3, analysis 3]; PR5I minus INFANRIX™ hexa

4. Primary Outcome: Percentage of Participants Vaccinated With PR5I Compared With INFANRIX™ Hexa With Acceptable Ab Response Rates to Hepatitis B and Seroresponse to Pertussis Antigens Pt, FHA and PRN One Month After the Toddler Dose at 13 Months Old
Description: Antibody titres were measured by ECi for HBsAg and ELISA for PT, FHA, & PRN. Percentage of participants with an Ab titre ≥10 mIU/mL HBsAg; ≥8 (1/dil) for IPV1, 2 & 3, and seroresponse to PT, FHA, and PRN are reported. The estimated response rates are based on the method by Miettinen and Nurminen stratified by country.
Time Frame: One month after Toddler dose of PRI5 (13 months old)
Population: All participants who met inclusion criteria, were not protocol violators, received vaccinations within acceptable day ranges, and who had serology results within RW of Days 28 to 51 Post-Toddler dose. Participants from site 0048 were excluded.
Measure: Number; unit: Percentage of participants
Arm/Group | PR5I | INFANRIX™ Hexa
Number analyzed (Participants) | 551 | 531
Percentage of participants
  Anti-HBsAg ≥10 mIU/mL | 99.64 | 99.06
  Anti-PT seroresponse: number analyzed (Participants) | 543 | 523
  Anti-PT seroresponse | 99.82 | 98.49
  Anti-FHA seroresponse: number analyzed (Participants) | 542 | 524
  Anti-FHA seroresponse | 97.22 | 99.81
  Anti-PRN seroresponse: number analyzed (Participants) | 543 | 523
  Anti-PRN seroresponse | 98.89 | 98.86
Statistical Analysis 1: Comparison: PR5I vs INFANRIX™ Hexa; Difference in percentages: Non-inferiority for HBsAg; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; p < 0.001, Miettinen & Nurminen — 1-sided; Difference in percentages = 0.58, 95% CI 2-sided [-0.49 to 1.85] — [estimate comment as in outcome 3, analysis 1]; PR5I minus INFANRIX™ hexa
Statistical Analysis 2: Comparison: PR5I vs INFANRIX™ Hexa; Difference in percentages: Non-inferiority for PT; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; p < 0.001, Miettinen & Nurminen — 1-sided; Difference in percentages = 1.33, 95% CI 2-sided [0.32 to 2.86] — [estimate comment as in outcome 3, analysis 1]; PR5I minus INFANRIX™ hexa
Statistical Analysis 3: Comparison: PR5I vs INFANRIX™ Hexa; Difference in percentages: Non-inferiority for FHA; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; p < 0.001, Miettinen & Nurminen — 1-sided; Difference in percentages = -2.59, 95% CI 2-sided [-4.39 to -1.29] — [estimate comment as in outcome 3, analysis 1]; PR5I minus INFANRIX™ hexa
Statistical Analysis 4: Comparison: PR5I vs INFANRIX™ Hexa; Difference in percentages: Non-inferiority for PRN; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; p < 0.001, Miettinen & Nurminen — 1-sided; Difference in percentages = 0.03, 95% CI 2-sided [-1.4 to 1.52] — [estimate comment as in outcome 3, analysis 1]; PR5I minus INFANRIX™ hexa

5. Secondary Outcome: Percentage of Participants Vaccinated With PR5I With Acceptable Ab Response to Measles, Mumps, Rubella and Varicella One Month After the Toddler Dose of ProQuad at 13 Months Old
Description: Ab titres were measured by ELISA, excepting the Ab to varicella which was determined by glycoprotein ELISA. Percentage of participants with an Ab titre ≥255 mIU/mL for measles, ≥10 Ab units/mL for mumps, ≥10 IU/mL for rubella, and ≥5 gpELISA units/mL for varicella are reported. 95% CI were calculated based on the exact binomial method by Clopper and Pearson. The immune response to ProQuad vaccine was considered as acceptable if the lower bounds of the 2-sided 95% CI for the response rates were greater than the predetermined lower CI limits: 90% for measles, mumps & rubella, and 76% for varicella.
Time Frame: One month after Toddler dose of PRI5 (13 months old)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PR5I
Number analyzed (Participants) | 467
Percentage of participants
  Anti-Measles ≥255 mIU/mL | 96.15 [93.98 to 97.7]
  Anti-Mumps ≥10 Ab units/mL | 94.86 [92.45 to 96.68]
  Anti-Rubella ≥10 IU/mL | 98.29 [96.65 to 99.26]
  Anti-Varicella ≥5 gpELISA units/mL | 97.64 [95.82 to 98.82]

6. Secondary Outcome: Percentage of Participants Vaccinated With PR5I Compared With INFANRIX™ Hexa With Acceptable Ab Response to Measles, Mumps, Rubella and Varicella One Month After the Toddler Dose of ProQuad at 13 Months Old
Description: Ab titres were measured by ELISA, excepting the Ab to varicella which was determined by glycoprotein ELISA. Percentage of participants with an Ab titre ≥255 mIU/mL for measles, ≥10 Ab units/mL for mumps, ≥10 IU/mL for rubella, and ≥5 gpELISA units/mL for varicella are reported. The estimated response rates are based on the method by Miettinen and Nurminen stratified by country.
Time Frame: One month after Toddler dose of PRI5 (13 months old)
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | PR5I | INFANRIX™ Hexa
Number analyzed (Participants) | 467 | 474
Percentage of participants
  Anti-Measles ≥255 mIU/mL | 96.15 | 96.41
  Anti-Mumps ≥10 Ab units/mL | 94.86 | 91.78
  Anti-Rubella ≥10 IU/mL | 98.28 | 97.89
  Anti-Varicella ≥5 gpELISA units/mL: number analyzed (Participants) | 467 | 471
  Anti-Varicella ≥5 gpELISA units/mL | 97.64 | 97.66
Statistical Analysis 1: Comparison: PR5I vs INFANRIX™ Hexa; Difference in percentages: Non-inferiority for Measles; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 3]; p < 0.001, Miettinen & Nurminen — 1-sided; Difference in percentages = -0.26, 95% CI 2-sided [-2.82 to 2.25] — [estimate comment as in outcome 3, analysis 3]; PR5I minus INFANRIX™ hexa
Statistical Analysis 2: Comparison: PR5I vs INFANRIX™ Hexa; Difference in percentages: Non-inferiority for Mumps; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 3]; p < 0.001, Miettinen & Nurminen — 1-sided; Difference in percentages = 3.07, 95% CI 2-sided [-0.12 to 6.4] — [estimate comment as in outcome 3, analysis 3]; PR5I minus INFANRIX™ hexa
Statistical Analysis 3: Comparison: PR5I vs INFANRIX™ Hexa; Difference in percentages: Non-inferiority for Rubella; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 3]; p < 0.001, Miettinen & Nurminen — 1-sided; Difference in percentages = 0.39, 95% CI 2-sided [-1.5 to 2.34] — [estimate comment as in outcome 3, analysis 3]; PR5I minus INFANRIX™ hexa
Statistical Analysis 4: Comparison: PR5I vs INFANRIX™ Hexa; Difference in percentages: Non-inferiority for Varicella; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; p < 0.001, Miettinen & Nurminen — 1-sided; Difference in percentages = -0.02, 95% CI 2-sided [-2.11 to 2.06] — [estimate comment as in outcome 3, analysis 1]; PR5I minus INFANRIX™ hexa

7. Secondary Outcome: Percentage of Participants With Injection-site and Systemic Adverse Events (AEs) From Day 1 to Day 15 After Any Vaccination
Description: Global safety was assessed by measuring injection-site and systemic AEs reported daily on the Vaccination Report Card (VRC) by the parent(s) or legal representative from Day 1 to Day 15 (D1-D15) after each hexavalent vaccination. Solicited injection-site and systemic AEs were reported daily from Day 1 to Day 5 (D1-D5) after each hexavalent vaccination. AEs at injection sites were always considered as vaccine-related (Injection-Site Reactions (ISRs)). The investigator assessed whether systemic AEs were related (V-related) or not to the vaccine. All AEs (related and unrelated) are reported.
Time Frame: Day 1 to Day 15 after any vaccination
Population: All randomised participants who received at least 1 vaccination and who had safety follow-up. Participants from site 0048 were excluded.
Measure: Number; unit: Percentage of participants
Arm/Group | PR5I | INFANRIX™ Hexa
Number analyzed (Participants) | 610 | 603
Percentage of participants
  At least 1 ISR or systemic AE (D1-D15) | 98.9 | 99.5
  At least 1 ISR or V-related systemic AE (D1-D15) | 98.5 | 98.8
  At least 1 ISR (D1-D15) | 92.1 | 91.0
  At least 1 solicited ISR (D1-D5): number analyzed (Participants) | 610 | 471
  At least 1 solicited ISR (D1-D5) | 90.8 | 89.9
  At least 1 systemic AE (D1-D15) | 98.4 | 99.3
  At least 1 V-related systemic AE (D1-D15) | 95.6 | 96.5
  At least 1 solicited systemic AE (D1-D5) | 97 | 98.5
  At least 1 V-related solicited systemic AE (D1-D5) | 94.9 | 96.2
Statistical Analysis 1: Comparison: PR5I vs INFANRIX™ Hexa; Risk difference: ISRs or systemic AEs; Test type: Other — Miettinen & Nurminen method; Risk Difference (RD) = -0.7, 95% CI 2-sided [-1.9 to 0.4] — If the 95% CI for the risk differences included 0.0, the numerical differences were not considered significant; PR5I minus INFANRIX™ hexa
Statistical Analysis 2: Comparison: PR5I vs INFANRIX™ Hexa; Risk difference: ISRs or vaccine-related systemic AEs; Test type: Other — Miettinen & Nurminen method; Risk Difference (RD) = -0.3, 95% CI 2-sided [-1.8 to 1.1] — If the 95% CI for the risk differences included 0.0, the numerical differences were not considered significant; PR5I minus INFANRIX™ hexa
Statistical Analysis 3: Comparison: PR5I vs INFANRIX™ Hexa; Risk difference: At least 1 ISR; Test type: Other — Miettinen & Nurminen method; Risk Difference (RD) = 1.1, 95% CI 2-sided [-2.1 to 4.3] — If the 95% CI for the risk differences included 0.0, the numerical differences were not considered significant; PR5I minus INFANRIX™ hexa
Statistical Analysis 4: Comparison: PR5I vs INFANRIX™ Hexa; Risk difference: At least 1 solicited ISR; Test type: Other — Miettinen & Nurminen method; Risk Difference (RD) = 0.9, 95% CI 2-sided [-2.4 to 4.3] — If the 95% CI for the risk differences included 0.0, the numerical differences were not considered significant; PR5I minus INFANRIX™ hexa
Statistical Analysis 5: Comparison: PR5I vs INFANRIX™ Hexa; Risk difference: At least 1 systemic AE; Test type: Other — Miettinen & Nurminen method; Risk Difference (RD) = -1, 95% CI 2-sided [-2.4 to 0.3] — If the 95% CI for the risk differences included 0.0, the numerical differences were not considered significant; PR5I minus INFANRIX™ hexa
Statistical Analysis 6: Comparison: PR5I vs INFANRIX™ Hexa; Risk difference: At least 1 vaccine-related systemic AE; Test type: Other — Miettinen & Nurminen method; Risk Difference (RD) = -0.9, 95% CI 2-sided [-3.2 to 1.3] — If the 95% CI for the risk differences included 0.0, the numerical differences were not considered significant; PR5I minus INFANRIX™ hexa
Statistical Analysis 7: Comparison: PR5I vs INFANRIX™ Hexa; Risk difference: At least 1 solicited systemic AE; Test type: Other — Miettinen & Nurminen method; Risk Difference (RD) = -1.5, 95% CI 2-sided [-3.3 to 0.2] — If the 95% CI for the risk differences included 0.0, the numerical differences were not considered significant; PR5I minus INFANRIX™ hexa
Statistical Analysis 8: Comparison: PR5I vs INFANRIX™ Hexa; Risk difference: At least 1 vaccine-related solicited systemic AE; Test type: Other — Miettinen & Nurminen method; Risk Difference (RD) = -1.3, 95% CI 2-sided [-3.7 to 1.1] — If the 95% CI for the risk differences included 0.0, the numerical differences were not considered significant; PR5I minus INFANRIX™ hexa

8. Secondary Outcome: Percentage of Participants Reporting Solicited ISRs From Day 1 to Day 5 After Any Vaccination
Description: Solicited ISRs were defined as injection-site erythema, injection-site pain, and injection-site swelling occurring from Day 1 (D1) to Day 5 (D5) after vaccination. AEs at injection sites were always considered as vaccine-related (Injection-Site Reactions (ISRs)).
Time Frame: Day 1 to Day 5 after any vaccination
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | PR5I | INFANRIX™ Hexa
Number analyzed (Participants) | 610 | 603
Percentage of participants
  Injection-site erythema | 69 | 64.2
  Injection-site pain | 73.6 | 71.8
  Injection-site swelling | 56.9 | 52.9
Statistical Analysis 1: Comparison: PR5I vs INFANRIX™ Hexa; Risk difference: Injection-site erythema; Test type: Other — Miettinen & Nurminen method; Risk Difference (RD) = 4.8, 95% CI 2-sided [-0.5 to 10.1] — If the 95% CI for the risk differences included 0.0, the numerical differences were not considered significant; PR5I minus INFANRIX™ hexa
Statistical Analysis 2: Comparison: PR5I vs INFANRIX™ Hexa; Risk difference: Injection-site pain; Test type: Other — Miettinen & Nurminen method; Risk Difference (RD) = 1.8, 95% CI 2-sided [-3.2 to 6.8] — If the 95% CI for the risk differences included 0.0, the numerical differences were not considered significant; PR5I minus INFANRIX™ hexa
Statistical Analysis 3: Comparison: PR5I vs INFANRIX™ Hexa; Risk difference: Injection-site swelling; Test type: Other — Miettinen & Nurminen method; Risk Difference (RD) = 4, 95% CI 2-sided [-1.6 to 9.6] — If the 95% CI for the risk differences included 0.0, the numerical differences were not considered significant; PR5I minus INFANRIX™ hexa

9. Secondary Outcome: Percentage of Participants Reporting Unsolicited ISRs From Day 1 to Day 15 After Any Vaccination
Description: Unsolicited ISRs with incidence ≥1% after any vaccination were reported daily on the VRC by the parent(s) or legal representative from (D1-D15). AEs at injection sites were always considered as vaccine-related ISRs
Time Frame: Day 1 to Day 15 after any vaccination
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | PR5I | INFANRIX™ Hexa
Number analyzed (Participants) | 610 | 603
Percentage of participants
  Injection-site bruising | 2.8 | 2.7
  Injection-site haematoma | 1.5 | 0.8
  Injection-site haemorrhage | 1.3 | 2.0
  Injection-site induration: number analyzed (Participants) | 610 | 471
  Injection-site induration | 14.6 | 18.2
  Injection-site nodule | 1.3 | 1.5
  Injection-site warmth | 3.0 | 1.8
Statistical Analysis 1: Comparison: PR5I vs INFANRIX™ Hexa; Risk difference: Injection-site bruising; Test type: Other — Miettinen & Nurminen method; Risk Difference (RD) = 0.1, 95% CI 2-sided [-1.8 to 2.1] — If the 95% CI for the risk differences included 0.0, the numerical differences were not considered significant; PR5I minus INFANRIX™ hexa
Statistical Analysis 2: Comparison: PR5I vs INFANRIX™ Hexa; Risk difference: Injection-site haematoma; Test type: Other — Miettinen & Nurminen method; Risk Difference (RD) = 0.6, 95% CI 2-sided [-0.6 to 2.1] — If the 95% CI for the risk differences included 0.0, the numerical differences were not considered significant; PR5I minus INFANRIX™ hexa
Statistical Analysis 3: Comparison: PR5I vs INFANRIX™ Hexa; Risk difference: Injection-site haemorrhage; Test type: Other — Miettinen & Nurminen method; Risk Difference (RD) = -0.7, 95% CI 2-sided [-2.3 to 0.8] — If the 95% CI for the risk differences included 0.0, the numerical differences were not considered significant; PR5I minus INFANRIX™ hexa
Statistical Analysis 4: Comparison: PR5I vs INFANRIX™ Hexa; Risk difference: Injection-site induration; Test type: Other — Miettinen & Nurminen method; Risk Difference (RD) = -3.7, 95% CI 2-sided [-7.8 to 0.5] — If the 95% CI for the risk differences included 0.0, the numerical differences were not considered significant; PR5I minus INFANRIX™ hexa
Statistical Analysis 5: Comparison: PR5I vs INFANRIX™ Hexa; Risk difference: Injection-site nodule; Test type: Other — Miettinen & Nurminen method; Risk Difference (RD) = -0.2, 95% CI 2-sided [-1.7 to 1.3] — If the 95% CI for the risk differences included 0.0, the numerical differences were not considered significant; PR5I minus INFANRIX™ hexa
Statistical Analysis 6: Comparison: PR5I vs INFANRIX™ Hexa; Risk difference: Injection-site warmth; Test type: Other — Miettinen & Nurminen method; Risk Difference (RD) = 1.1, 95% CI [-0.6 to 3] — If the 95% CI for the risk differences included 0.0, the numerical differences were not considered significant; PR5I minus INFANRIX™ hexa

10. Secondary Outcome: Percentage of Participants Reporting Solicited Systemic AE From Day 1 to Day 5 After Any Vaccination
Description: Solicited systemic AEs were defined as crying, decreased appetite, irritability, pyrexia (rectal temperature ≥38.0°C), somnolence, and vomiting occurring from D1 to D5 after vaccination. The investigator assessed whether these systemic AEs were related or not to the vaccines. All (related and unrelated) AEs are reported.
Time Frame: Day 1 to Day 5 after any vaccination
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | PR5I | INFANRIX™ Hexa
Number analyzed (Participants) | 610 | 603
Percentage of participants
  Crying | 85.4 | 87.9
  Decreased appetite | 63.9 | 67.0
  Irritability | 87.9 | 85.7
  Pyrexia | 71.5 | 73.1
  Somnolence | 76.9 | 80.1
  Vomiting | 31.8 | 31.0
Statistical Analysis 1: Comparison: PR5I vs INFANRIX™ Hexa; Risk difference: Crying; Test type: Other — Miettinen & Nurminen method; Risk Difference (RD) = -2.5, 95% CI 2-sided [-6.3 to 1.4] — If the 95% CI for the risk differences included 0.0, the numerical differences were not considered significant; PR5I minus INFANRIX™ hexa
Statistical Analysis 2: Comparison: PR5I vs INFANRIX™ Hexa; Risk difference: Decreased appetite; Test type: Other — Miettinen & Nurminen method; Risk Difference (RD) = -3.1, 95% CI 2-sided [-8.4 to 2.3] — If the 95% CI for the risk differences included 0.0, the numerical differences were not considered significant; PR5I minus INFANRIX™ hexa
Statistical Analysis 3: Comparison: PR5I vs INFANRIX™ Hexa; Risk difference: Irritability; Test type: Other — Miettinen & Nurminen method; Risk Difference (RD) = 2.1, 95% CI 2-sided [-1.7 to 6] — If the 95% CI for the risk differences included 0.0, the numerical differences were not considered significant; PR5I minus INFANRIX™ hexa
Statistical Analysis 4: Comparison: PR5I vs INFANRIX™ Hexa; Risk difference: Pyrexia; Test type: Other — Miettinen & Nurminen method; Risk Difference (RD) = -1.7, 95% CI 2-sided [-6.7 to 3.4] — If the 95% CI for the risk differences included 0.0, the numerical differences were not considered significant; PR5I minus INFANRIX™ hexa
Statistical Analysis 5: Comparison: PR5I vs INFANRIX™ Hexa; Risk difference: Somnolence; Test type: Other — Miettinen & Nurminen method; Risk Difference (RD) = -3.2, 95% CI 2-sided [-7.8 to 1.4] — If the 95% CI for the risk differences included 0.0, the numerical differences were not considered significant; PR5I minus INFANRIX™ hexa
Statistical Analysis 6: Comparison: PR5I vs INFANRIX™ Hexa; Risk difference: Vomiting; Test type: Other — Miettinen & Nurminen method; Risk Difference (RD) = 0.8, 95% CI 2-sided [-4.4 to 6] — If the 95% CI for the risk differences included 0.0, the numerical differences were not considered significant; PR5I minus INFANRIX™ hexa

ADVERSE EVENTS:
Time Frame: 2 months after Toddler Dose (up to approximately age 14 months)
Description: All Treated Participants. Participants from site 0048 were excluded.
Groups:
- INFANRIX Hexa: The INFANRIX™ hexa group received INFANRIX™ hexa, Prevenar 13™, and RotaTeq™ at 2, 3, and 4 months; followed by INFANRIX™ hexa and ProQuad™ at 12 months; and Prevenar 13™ and ProQuad™ at 13 months.
Arm/Group | PR5I | INFANRIX Hexa
All-Cause Mortality (participants affected / at risk) | 0/610 | 0/605
Serious Adverse Events (participants affected / at risk) | 23/610 | 22/605
Other Adverse Events (participants affected / at risk) | 603/610 | 599/605
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PR5I (N=610) | INFANRIX Hexa (N=605)
Benign familial neonatal convulsions (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Swollen tongue (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 2 (2)
Bronchiolitis (Infections and infestations) | 3 (3) | 2 (2)
Bronchitis (Infections and infestations) | 2 (2) | 1 (1)
Bronchitis viral (Infections and infestations) | 0 (0) | 1 (1)
Exanthema subitum (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Pneumococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 2 (4) | 2 (2)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 3 (3) | 7 (7)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Abdominal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Prolymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Febrile convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Neuroendocrine cell hyperplasia of infancy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PR5I (N=610) | INFANRIX Hexa (N=605)
Conjunctivitis (Eye disorders) | 20 (23) | 32 (36)
Diarrhoea (Gastrointestinal disorders) | 98 (129) | 84 (113)
Flatulence (Gastrointestinal disorders) | 45 (55) | 39 (50)
Vomiting (Gastrointestinal disorders) | 205 (328) | 194 (333)
Crying (General disorders) | 523 (1543) | 531 (1482)
Injection site erythema (General disorders) | 459 (1745) | 430 (1517)
Injection site induration (General disorders) | 106 (245) | 127 (296)
Injection site pain (General disorders) | 469 (1710) | 456 (1637)
Injection site swelling (General disorders) | 384 (1214) | 347 (1101)
Irritability (General disorders) | 537 (1639) | 518 (1570)
Pyrexia (General disorders) | 471 (1072) | 472 (1065)
Nasopharyngitis (Infections and infestations) | 24 (29) | 35 (41)
Otitis media (Infections and infestations) | 32 (33) | 26 (30)
Rhinitis (Infections and infestations) | 82 (102) | 86 (101)
Upper respiratory tract infection (Infections and infestations) | 69 (82) | 76 (83)
Decreased appetite (Metabolism and nutrition disorders) | 401 (752) | 408 (718)
Somnolence (Nervous system disorders) | 470 (1082) | 485 (1058)
Cough (Respiratory, thoracic and mediastinal disorders) | 35 (39) | 38 (44)
Rash (Skin and subcutaneous tissue disorders) | 35 (42) | 27 (32)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR and SPONSOR representative must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR or SPONSOR representative as confidential must be deleted prior to submission.